CLINICAL TRIAL: NCT04758871
Title: Dydrogesterone Versus Micronized Vaginal Progesterone (MVP) for Luteal Phase Support (LPS) in Hormone Replacement Therapy (HRT) Frozen Embryo Transfer (FET) Cycles.
Brief Title: Oral Versus Vaginal Progesterone for Luteal Phase Supplementation in Frozen Embryo Transfer Cycles
Acronym: REMODEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CRG UZ Brussel (Other)
Responsible Party: Principal Investigator, Caroline Roelens, Co-investigator, CRG UZ Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMODEL
Record Dates: First submitted 2021-01-26; First posted 2021-02-17 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Frozen Embryo Transfer; Hormone Replacement Therapy; Dydrogesterone; Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Dydrogesterone; Tablets; Progesterone

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dydrogesterone (Experimental): Luteal phase support for hormone replacement therapy frozen embryo transfer cycles using dydrogesterone 10 mg 3 times daily
  Interventions: Drug: Dydrogesterone 10 MG Oral Tablet
- Micronized progesterone (Active Comparator): Luteal phase support for hormone replacement therapy frozen embryo transfer cycles using micronized progesterone 2x200 mg twice daily vaginally
  Interventions: Drug: Micronized progesterone

INTERVENTIONS:
Drug: Dydrogesterone 10 MG Oral Tablet — 10 mg three times daily
  Arms: Dydrogesterone
Drug: Micronized progesterone — 2x 200 mg vaginal tablets two times daily
  Arms: Micronized progesterone

SUMMARY:
To investigate the efficacy of dydrogesterone 30 mg compared to micronized vaginal progesterone 800 mg daily for luteal phase support in hormone replacement therapy frozen embryo transfer cycles, as confirmed by visualization of fetal heart activity by pelvic ultrasound assessment of ongoing pregnancy at 12 weeks of gestation.

DETAILED DESCRIPTION:
A randomized controlled trial comparing dydrogesterone 30 mg versus micronized vaginal progesterone 800 mg daily for luteal phase support in hormone replacement therapy frozen embryo transfer cycles. Patients will undergo an embryo transfer in a hormone replacement therapy cycle using Progynova 2 mg three times daily until an endometrium thickness of at least 7 mm is reached. Afterwards two different luteal phase supplementation methods will be compared. The primary outcome of the study is ongoing pregnancy at 12 weeks of gestation. We will also investigate other prenatal and neonatal outcome factors as well as patients satisfaction and safety of dydrogesterone.

ELIGIBILITY:
Inclusion Criteria:

* ≤40 years of age at the time of IVF/ICSI treatment
* BMI ≥18 to ≤30 kg/m2 with a documented history of infertility
* Have undergone COS as part of an ART treatment and have had an unsuccessful fresh embryo transfer in that cycle, OR, have undergone freeze all strategy
* Scheduled to undergo FET with a standard exogenous/programmed hormonal replacement therapy (HRT) regimen
* Have at least 1 blastocyst vitrified on the 5th or 6th day after oocyte retrieval
* Elective single embryo (blastocyst) transfer (SET)
* Normal ultrasound examination at enrollment (or if <12 months old)
* Signed patient authorization for use/disclosure of data.

Exclusion Criteria:

* Women with a history of recurrent miscarriage, defined as >2 consecutive miscarriages (biochemical pregnancy losses are not included)
* Absence of implantation (serum hCG = negative) after two consecutive cycles of IVF, ICSI or FET where the cumulative number of transferred embryos was >4 cleavage-stage embryos and >2 blastocysts
* Presence of hydrosalpinx that is not surgically treated
* Endometrial abnormalities on scanning during ovarian stimulation, such as endometrial polyp(s), sub mucosal fibroid(s), endometrial hyperplasia, endometrial fluid accumulation, or endometrial adhesions
* Participating in another clinical study at the same time
* Known allergic reactions to dydrogesterone or other progestogens products
* Any contraindication or other condition that precludes use of dydrogesterone in a particular patient, in accordance with the precautions listed in the locally approved label
* Mental disability or any other lack of fitness, in the Investigator's opinion, to preclude subjects in or to complete the study
* History of prior chemotherapy
* Contraindication for pregnancy
* Transfer of >1 embryo

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy | 12 weeks
  visualisation of a fetal heart activity via pelvic (vaginal/abdominal) ultrasound examination at 12 weeks of gestation.

SECONDARY OUTCOMES:
Live birth rate | 22-42 weeks
  as the birth of a live newborn after 22 weeks of gestation
Time of delivery | follow-up time of 30 days after delivery
  time of delivery (gestational week) will be confirmed (by calculation from date of embryo transfer)
Incidence of Treatment-Emergent Adverse Events | follow-up time of 30 days after delivery
  Tolerability and safety will be asses during the whole study period. Adverse events will be considered as unexpected if the nature, seriousness, severity or outcome of the reaction(s) is not consistent with the reference information. The expectedness of adverse events for the medications used in this study is detailed in the reference safety information in the current summary of product characteristics (SmPCs) issued in the participating countries.
  All serieus suspected unexpected serious adverse drug reactions (SUSARs) will be subject to expedited reporting. The investigator is responsible for submitting reports of SUSARs to the appropriate national regulatory authorities within the required reporting period. The investigator is responsible for notifying the IECs/IRBs in writing of the SUSARs within the required reporting timelines. Copies of the notification will be maintained by the investigator in the study documentation files.
Patient reported outcome | day 12-18 of luteal phase supplementation (pregnancy test) and at 12 weeks gestation
  Questionnaire (using the Treatment Satisfaction Questionnaire of Medication (TSQM)) and recording information on treatment tolerability and convenience
Incidence of newborn adverse events | follow-up time of 30 days after delivery
  Newborn wellbeing and safety including congenital malformations will be evaluated after delivery via a telephonic contact with the patient
Biochemical pregnancy rate | day 12-18 of luteal phase supplementation (pregnancy test)
  serum hCG test (> 25 mIU/ml), without ultrasound evaluation of a pregnancy
Clinical pregnancy rate | Day 33-39 of LPS (Verification of pregnancy)
  assessed by transvaginal ultrasound and defined as the presence of ≥1 gestational sac on examination
Miscarriage rate | 22 weeks
  defined as spontaneous loss of a clinical pregnancy before 22 weeks of gestation (where embryo(s) or fetus(es) is/are nonviable and is/are not spontaneously absorbed or expelled from the uterus)
Rate of preterm birth | follow-up time of 30 days after delivery
  Delivery before 37 weeks of gestation
Rate of pre-eclampsia | follow-up time of 30 days after delivery
  Incidence of pre-eclampsia as defined by the defined as the development of hypertension after 20 weeks of gestation together with one or more new-onset conditions: proteinuria, maternal or uteroplacental dysfunctions. Univariate and multivariable regression analysis were performed to control for known or potential PE risk factors, more specifically: body mass index (BMI), African ethnicity, previous history of hypertensive disorders of pregnancy, mean arterial pressure (MAP) at the first prenatal consultation, polycystic ovary syndrome (PCOS) and ovulation disorders, endometrial thickness and oocyte recipients.
Occurence of antenatal bleeding, ultrasonographic abnormalities, gestational diabetes, cholestasis | follow-up time of 30 days after delivery
  Occurence of antenatal bleeding, ultrasonographic abnormalities, gestational diabetes, cholestasis
Implantation rate | Day 33-39 of LPS (Verification of pregnancy)
  assessed by ultrasound and defined as the number of gestational sacs per number of embryos transferred
Blastocyst development score | at the time of embryo transfer (visit 2: day 6 of luteal phase supplementation)
  using the system developed by Gardner
Number of cryopreserved embryos | day of screening and enrollment
  Number of cryopreserved embryos
Summary characteristics of the preceding controlled ovarian stimulation cycle | day of screening and enrollment
  information on used stimulation medication, total dose of stimulation medication used, duration of stimulation medication, trigger medication

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Blockeel, Principal Investigator — CRG UZ Brussel
Locations (1):
- Brussels IVF, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No